CLINICAL TRIAL: NCT07027514
Title: A Phase 1b, Two-Part Study of Tolododekin Alfa (ANK-101) in Combination With an Anti-PD-1/PD-L1 Antibody in Participants With Advanced Non-Small Cell Lung Cancer
Brief Title: A Study of Tolododekin Alfa (ANK-101) in Combination With an Anti-PD-1/PD-L1 Antibody in Participants With Advanced Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ankyra Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANK-101-004
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Participants will receive up to 8 cycles of tolododekin alfa in combination with cetrelimab given for up to 1 year
  Interventions: Drug: tolododekin alfa; Drug: Cetrelimab
- Cohort B (Experimental): Participants will receive up to 8 cycles of tolododekin alfa in combination with the Investigator's choice of a Food and Drug Administration (FDA)-approved anti-PD-1/PD-L1 antibody given according to the FDA-approved label
  Interventions: Drug: tolododekin alfa

INTERVENTIONS:
Drug: tolododekin alfa — Participants will receive tolododekin alfa as an intratumoral injection every 3 weeks (Q3W).
Drug: Cetrelimab — Participants will receive cetrelimab Q3W.
  Arms: Cohort A

SUMMARY:
A study of tolododekin alfa (also known as ANK-101) administered in combination with an anti-programmed cell death protein 1 (PD-1)/programmed cell death ligand 1 (PD-L1) antibody in participants with advanced or metastatic non-small cell lung cancer (NSCLC). Cohort A will enroll participants who have progressed on prior standard of care treatment with an anti-PD-1/PD-L1 antibody and a platinum-based chemotherapy regimen. Cohort B will enroll participants who are treatment-naïve for locally advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Have confirmed locally advanced or metastatic NSCLC
2. Thyroid-stimulating hormone (TSH) within normal limits
3. Have measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
4. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 to 1
5. Have a life expectancy > 12 weeks
6. Have baseline electrocardiogram (ECG) without evidence of acute ischemia or prolonged QT interval
7. Heterosexually active women of childbearing potential (WOCBP) must agree to use at least 2 forms of highly effective methods of contraception
8. All male participants who are not sterile must commit to the use of a reliable method of birth control or abstinence
9. Human immunodeficiency virus (HIV)-infected participants must be on anti-retroviral therapy (ART) and have well-controlled HIV infection/disease
10. Resolution of all prior anticancer therapy toxicities to ≤ Grade 1 prior to C1D1.
11. Willingness to provide fresh tumor biopsy specimens
12. Capable of understanding and complying with protocol requirements
13. Provides written informed consent for the study

Exclusion Criteria:

1. Cohort A only: Participants with Grade 3 or higher toxic effects to manage adverse events from previous treatment with immunotherapy
2. Cohort B only: Prior therapy with an immune checkpoint inhibitor.
3. Have known EGFR or ALK mutations
4. Have had prior treatment with recombinant interleukin-12 (IL-12)
5. Have received short-term systemic therapy with immunosuppressive agents prior to C1D1
6. Have active autoimmune disease or medical conditions requiring chronic steroid or other immunosuppressive therapy prior toC1D1
7. Have received live vaccines within 28 days prior to C1D1
8. Have primary or acquired immunodeficient states
9. Women of childbearing potential who has a positive serum pregnancy test prior to C1D1 or female participant who is breastfeeding
10. Have a history of allogeneic tissue/solid organ transplant
11. Has known active uncontrolled hepatitis B virus (HBV) or hepatitis C virus (HCV).
12. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease
13. Have known active central nervous system metastases
14. Have congestive heart failure, active coronary artery disease, unevaluated new onset angina, unstable angina, or clinically significant cardiac arrhythmias.
15. Have uncontrolled bleeding disorders prior to C1D1
16. Participants on coumadin (warfarin), due to potential for increased bleeding risk associated with surgery
17. History of noninfectious pneumonitis within the previous 5 years
18. Cohort A only: History of allergy to protein-based therapies, history of any significant drug allergy, or known allergies, hypersensitivity, or intolerance to cetrelimab excipients OR Cohort B only: Hypersensitivity to any component of the anti-PD-1/PD-L1 antibody selected as standard of care
19. Have other systemic conditions or organ abnormalities that may interfere with the conduct of the study
20. Have any acute or chronic psychiatric problems or substance abuse disorder that make the participant unsuitable for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 | 6 months
  Percentage of participants with complete response (CR) or partial response (PR) among all response evaluable participants

SECONDARY OUTCOMES:
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | 6 months
  Number of participants with adverse events (TEAEs, SAEs)
Duration of Response (DoR) | 6 months
  Time from first CR/PR to the date of progressive disease (PD) or death.
Disease Control Rate (DCR) | 6 months
  The percentage of participants with stable disease, complete response or partial response among all response evaluable participants
Progression Free Survival (PFS) | 6 months
  The duration from the first dose of tolododekin alfa until PD/death
Overall Survival (OS) | 6 months
  The length of time participants remain alive starting from the first dose of tolododekin alfa
Lesion-level response in injected and noninjected lesions | 6 months
  Measure response in injected and noninjected lesions
Measure of area under the plasma concentration-time curve (AUC) of tolododekin alfa | 6 months
  Characterize pharmacokinetic (PK) parameter AUC after IT injection of tolododekin alfa
Measure of maximum plasma concentration (Cmax) of tolododekin alfa | 6 months
  Characterize pharmacokinetic (PK) parameter Cmax after IT injection of tolododekin alfa
Measure of time to maximum concentration (Tmax) of tolododekin alfa | 6 months
  Characterize pharmacokinetic (PK) parameter Tmax after IT injection of tolododekin alfa
Measure of volume of distribution adjusted for bioavailability (Vd/F) of tolododekin alfa | 6 months
  Characterize pharmacokinetic (PK) parameter Vd/F after IT administration of tolododekin alfa
Measure of terminal half-life (t1/2) of tolododekin alfa | 6 months
  Characterize pharmacokinetic (PK) parameter t1/2 after IT administration of tolododekin alfa
Incidence of treatment-emergent anti-drug antibodies (ADA) of tolododekin alfa | 6 months
  Quantification of ADAs after IT administration of tolododekin alfa

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Community Health Network, Indianapolis, Indiana
  - Barbara Ann Karmanos Cancer Hospital, Detroit, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - FirstHealth of the Carolinas, Pinehurst, North Carolina

IPD SHARING:
Plan to Share IPD: No